CLINICAL TRIAL: NCT02398890
Title: Follow-up of Oncology Patients After Hospitalization in ICU
Acronym: SALTO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: KI120906; 2013-A00683-42 (Other: ANSM)
Record Dates: First submitted 2014-12-19; First posted 2015-03-26 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2018-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: routine care — routine care

SUMMARY:
"Purpose: The overall prognosis of oncology patients admitted to intensive care has improved greatly in recent years, leading to a wider admission policy. Due to a decrease in mortality in intensive care, more and more patients returning oncological circuit for the continuation of treatment of the underlying disease The existence of sequelae after the ICU (Intensive Care Unit) stay, whether renal, cardiac, respiratory or other, may influence the continuation of the optimal anti -cancer treatments and thus reduce the chances of recovery or evolution without tumor progression. However, no studies have evaluated the effects of resuscitation on subsequent cancer treatment strategies. It would thus become better appreciate the long-term oncology patients discharged alive from the hospital after a stay in intensive care.

Main purpose of research :

Assess the feasibility of a anti-tumor therapy for patients with progressive solid tumors, after an intensive care stay for other reason than elective surgery monitoring or securing an invasive procedure. The possibility of making an anti -cancer treatment will be evaluated by the treating oncologist and classified total, partial or absent from that defined before or during the ICU stay

Secondary objective of the research :

Evaluate the percentage of patients discharged alive from the ICU and dying in the hospital.

Evaluate survival, lifestyle and physical and psychological effects of these patients after discharge from the hospital over a period of one year. It is understood that all these secondary endpoints will interfere with the existence of an evolutionary neoplasia not only with the ICU stay. They will therefore be interpreted with caution.

Study Type: observational Study Design: Prognostic study of routine care, national, prospective, cohort type "

DETAILED DESCRIPTION:
"Nature of evaluated care: Longitudinal follow-up of post- resuscitation intensive care Concerned population: adult patients with active solid tumor out alive from the ICU and following-up in oncology in the same hospital as the resuscitator investigator.

Main objective: Measure the influence of ICU for patients with solid cancers to continue with optimal anti -cancer treatment, defined before or during hospitalization in intensive care.

Secondary objective: Assess the physical and psychological consequences of ICU stay of patients Evaluation criteria : Primary endpoint: proportion of patients living, out from ICU and hospital, can receive optimal cancer treatment later.

Research Methodology : Prognostic study of routine care, national, prospective, cohort type."

ELIGIBILITY:
Inclusion criteria:

* Patient with progressive solid tumor hospitalized in intensive care and got out alive
* Oncology patients followed in the same hospital as the investigator resuscitator
* Age ≥ 18 years
* Affiliate of social insurance
* Agree to participate

Exclusion criteria :

* Patient hospitalized for programed surgery
* Hospitalization for securing procedure
* Pregnancy or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with active solid tumor out alive from the ICU and monitoring in oncology in the same hospital as the resuscitator investigator.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with cancer admitted in ICU who will be eligible for optimal anti-cancer treatment after discharge from ICU | Months12

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Le Raincy-Montfermeil, Montfermeil, France